CLINICAL TRIAL: NCT03422523
Title: A Phase II Study of Atezolizumab With Rituximab, Gemcitabine and Oxaliplatin in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma Who Are Not Candidates for High-dose Therapy
Brief Title: Atezolizumab, Rituximab, Gemcitabine and Oxaliplatin in Patients With Relapsed or Refractory DLBCL Not Suitable for High-dose Therapy
Acronym: ARGO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to reach pre-specified futility boundary
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHM CAN1219; 2016-002654-21 (EudraCT Number)
Record Dates: First submitted 2018-01-11; First posted 2018-02-05 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Diffuse Large B Cell Lymphoma; Relapsed Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
Keywords: Refractory; Relapsed; Hematological cancer
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — atezolizumab; Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A Control (Active Comparator): 6 Cycles of R-GemOx (Rituximab, Gemcitabine and Oxaliplatin) every 14 days.
  Interventions: Drug: Rituximab; Drug: Gemcitabine 1000 mg; Drug: Oxaliplatin 100 MG
- Arm B Experimental (Experimental): 1 Cycle of R-GemOx (Rituximab, Gemcitabine and Oxaliplatin) followed by 5 cycles of R-GemOx with Atezolizumab every 14 days.
  Followed by 8 maintenance cycles of Atezolizumab every 21 days.
  Interventions: Drug: Atezolizumab; Drug: Rituximab; Drug: Gemcitabine 1000 mg; Drug: Oxaliplatin 100 MG

INTERVENTIONS:
Drug: Atezolizumab — Intravenous drip
  Other Names: Tecentriq
  Arms: Arm B Experimental
Drug: Rituximab — Intravenous drip/or Subcutaneous from cycle 2
  Other Names: Mabthera
Drug: Gemcitabine 1000 mg — intravenous drip
Drug: Oxaliplatin 100 MG — intravenous drip

SUMMARY:
This study evaluates the addition of Atezolizumab to current therapy of Rituximab, Gemcitabine and Oxaliplatin (R-GemOx) for patients with relapsed or refractory Diffuse Large B-Cell Lymphoma (DLBCL) that are not candidates for high-dose therapy. All patients will receive one cycle of R-GemOx. Three quarters of patients (Arm B) will go on to have a further 5 cycles (every 14 days) of R-GemOx with Atezolizumab, with one quarter of patients (Arm A) continuing with 5 cycles of R-GemOx.

The patients in Arm B will continue to have Atezolizumab every 21 days for 8 cycles whilst Arm A patients will enter an observational phase during this time.

Follow up will begin at 12 months from initial treatment until month 32.

DETAILED DESCRIPTION:
Rituximab is a chimeric mouse/human monoclonal antibody that binds to CD20, on pre-B and mature B lymphocytes and eliminates these cells potentially via a number of different mechanisms.

The R-GemOx regimen has been adopted by many sites internationally as therapy for older patients or comorbid patients with relapsed or refractory DLBCL and as a back-bone for the investigation of novel therapies in combination with chemotherapy.

The cytotoxic T-lymphocyte co-receptor PD-1 has been extensively studied and is recognised to provide critical inhibitory signals that down-regulate T-cell function and provides a mechanism for immune evasion for tumours. PD-L1, the ligand of PD-1 is expressed on DLBCL tumour cells, along with infiltrating non-malignant cells, primarily macrophages, with PD-1 expressed on tumour infiltrating lymphocytes (TILs). Atezolizumab targets programmed PD-L1 on immune and tumour cells and prevents interaction with either PD-1 receptor or B7.1 (CD80), both of which function as inhibitory receptors expressed on T cells. Interference of the PD-L1:PD-1 and PDL1:B7.1 interactions may enhance the magnitude and quality of the tumour-specific T-cell response through increased T-cell priming, expansion, and/or effector function.

This study of atezolizumab in combination with rituximab, gemcitabine and oxaliplatin aims to address the unmet need of patients with relapsed and refractory DLBCL. It is based upon a sound mechanistic approach, investigating the activity of novel agents and will aim to compressively explore biomarkers of response.

The primary objective will be to document the durability of anti-tumour activity in patients with relapsed or refractory DLBCL and to determine the safety and toxicity profile of the combination. A maintenance phase of atezolizumab has been added as this may induce an on-going T-cell response to neo-antigens released as a result of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CD20 +ve diffuse large B-cell lymphoma with sufficient diagnostic material, obtained either at diagnosis or relapse (the latter is preferable) that is available to forward to the Haematological Malignancies Diagnostic Service (HMDS) for gene expression profiling and central pathology review. (See screening procedure for details on biopsy requirements)
* Refractory to, or relapsed following, first-line or second-line treatments with rituximab concurrently with anthracycline or anthracenedione-based chemotherapy (etoposide or gemcitabine allowed if comorbid).

Refractory disease must fulfil one of the following:

* Continuing partial response (PR) from termination of first-line treatment. It is strongly recommended the lymphoma be reconfirmed by biopsy however, if these procedures are deemed to be inappropriate, the CI may determine eligibility following review of the imaging results and disease history.
* Continuing stable disease (SD) from termination of first-line treatment. Reconfirmation of the lymphoma by biopsy (preferred) is recommended but not mandatory.
* Progressive disease (PD). Biopsy or reconfirmation of the lymphoma is recommended but not mandatory.

  o Not eligible for high-dose therapy with peripheral blood progenitor cell rescue at Investigator discretion as a result of:
* Age
* Co-morbidity
* Previous HDT. Rationale to be clearly documented on eCRF and medical notes.

  * Baseline FDG-PET scans must demonstrate positive lesions compatible with CT defined anatomical tumour sites.
  * CT/PET scan showing at least:
* 2 or more clearly demarcated lesions/nodes with a long axis >1.5cm and short axis ≥1.0cm OR
* 1 clearly demarcated lesion/node with a long axis >2.0cm and short axis ≥1.0cm.

  * Resolution of toxicities from previous therapy to a grade that in the opinion of the investigator does not contraindicate study participation.
  * Patients aged 16 years or over.
  * Willingness to participate in appropriate pregnancy prevention measures.
* Female patients who are fertile and of childbearing potential must have a negative serum or urine pregnancy test during screening (within 14 days prior to the start of trial treatment) and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom; an intra-uterine device and condom) effective from the first administration of all study drugs, throughout the trial and for 12 months after last dose of study therapy are considered eligible. Unless they are surgically sterile or ≥ 2 years after the onset of menopause.
* Male patients with partners of child-bearing potential who agree to take measures not to father children by using one form of highly effective contraception (oral, injected or implanted hormonal contraception and condom; an intra-uterine device and condom) effective from the first administration of all study drugs, throughout the trial and for 12 months after last dose of study therapy are considered eligible. Male subjects must also refrain from donating sperm during this period. Unless they are surgically sterile.
* Men with pregnant or lactating partners must be advised to use barrier method contraception (for example: condom plus spermicidal gel) to prevent exposure to the foetus or neonate

  * Written informed consent using current version of Protocol, Patient Information Sheet and Informed Consent Form.
  * ECOG performance status ≤3

Exclusion Criteria:

* Received any of the following treatments within two weeks prior to start of study therapy (unless otherwise stated):

  * Anti-cancer cytotoxics (excluding corticosteroids)
  * Radiotherapy unless it is to a limited field to control life/organ-threatening symptoms.
* DLBCL that is refractory to or relapsed within 3 months of a gemcitabine regimen for DLBCL
* Major surgery within 4 weeks of registration.
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half-lives or 4 weeks prior to registration.
* History of stroke or intracranial haemorrhage within 6 months prior to registration.
* Pre-existing peripheral neuropathy grade >2.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to registration, congestive heart failure (NYHA III-IV), a current LVEF of <40%
* Significant concurrent, uncontrolled medical condition that in the opinion of the investigator contraindicates participation in this study
* Known lymphoma involvement of the CNS.
* Known or suspected hypersensitivity to study treatments that in the opinion of the investigator contraindicates their participation. Patients with known history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug induced pneumonitis or idiopathic pneumonitis, or evidence of active pneumonitis will be excluded from study participation.
* Known HIV positivity; positive serology for Hep B (defined as positivity for Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (anti-HBc)) or C; chronic or current infectious disease (except evidence of prior vaccination).
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 2 weeks of the start of Cycle 1. Suspected active or latent tuberculosis needs to be confirmed by positive interferon gamma (IFN-gamma) release assay.
* Other past or current malignancy within 2 years prior to registration unless in the opinion of the investigator it does not contraindicate participation in the study. Subjects who have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma, are eligible.
* Screening laboratory values:
* platelets <75x109/L (unless due to lymphoma involvement of the bone marrow)
* neutrophils <1.0x109/L (unless due to lymphoma involvement of the bone marrow)
* creatinine >2.0 times upper normal limit (unless due to lymphoma or unless creatinine clearance >60mL/min (should be calculated using Cockcroft and Gault equation))
* total bilirubin >1.5 times upper normal limit (unless due to lymphoma or a known history of Gilbert's disease, no higher than >3 times upper normal limit)
* ALT/AST >2.5 times upper normal limit (unless due to lymphoma, no higher than >5 times upper normal limit)
* alkaline phosphatase >2.5 times upper normal limit (unless due to lymphoma, no higher than >5 times upper normal limit)
* Subjects known or suspected of being unable to comply with the study protocol.
* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test at screening.
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis (Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone will be eligible as will be patients with controlled Type I diabetes mellitus on a stable dose of insulin). Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
* Rash must cover <10% of body surface area
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
* Patients who have previously undergone allogeneic transplantation.
* Vaccination with a live vaccine within 28 days of study treatment or anticipation of need for such a vaccine during the course of the study and up to 5 months after the last dose of atezolizumab.
* History of severe allergic anaphylactic reactions to chimeric, human or humanised antibodies, or fusion proteins.
* Known hypersensitivity to CHO cell products or any component of the atezolizumab formulation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Progression free survival | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, up to follow up at month 36.
  Progression free survival will be measured from patient notes, from the day of registration to the date of progression or death from any cause. Patients who do not die will be censored at their date of last follow up.

SECONDARY OUTCOMES:
AE's reported and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) for R-GemOx-Atezo | At all visits from baseline to follow up month 36
  Determining the toxicity and causality of each adverse event with R-GemOx-Atezo.
Lugano classification lymphoma response criteria (LYRIC) to PET/CT | Baseline and cycle 3 day 8, cycle 3 day 8 and week 42, week 42 and 12 month follow up, 12 month follow up and 24 month follow up
  Objective response, partial or complete metabolic response, to be assessed by PET / CT according to LYRIC.
Overall survival | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, up to follow up at month 36.
  Overall survival will be measured from patient notes, from the day of registration to the date of death from any cause. Patients who do not die will be censored at their date of last follow up.

OTHER OUTCOMES:
Whole transcriptome profiling | Baseline
  Gene expression profiling on FFPE tumour material
Double staining techniques | Baseline
  immunohistochemical analysis of primary tumour material
Flow Cytometry | day 1 of cycles 1, 2, 3, and 5, week 15, day 1 of weeks 17, 23, 29, 35 and 42 only
  flow cytometry of t-cells in peripheral blood collected during therapy
Genes of NGS DLBCL mutation panel | Baseline
  Application genes of NGS DLBCL mutation panel of 54 genes to tumour material
Fluorescence in situ Hybridization (FISH) analysis | Baseline
  Examine translocations of Myc, Bcl6 and Bcl2 by FISH
Immunohistochemical analysis for dual protein expression | Baseline
  Immunohistochemical analysis for dual protein expression on Myc and Bcl2
cfDNA molecular analysis | baseline, cycle 2 day 1, cycle 3 day 1, cycle 5 day 1, week 15, day 1 week 29, day 1 week 38 and follow up months 12, 16, 20, 24, 30 and 36.
  Plasma lymphoma nucleic acid at baseline studied and compared with paired lymphoma tissue sample and repeated throughout study period to examine dynamics of change and possible assessment of minimal residual disease, depending upon responses observed

CONTACTS AND LOCATIONS:
Overall Officials: Andy Davies, Principal Investigator — Southampton University
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided